CLINICAL TRIAL: NCT06586827
Title: The Impact of Competency-Based Training and Technical Assistance on the Competitive Integrated Employment Outcomes of Individuals With ID/DD
Brief Title: Impact of Competency-Based Training and Technical Assistance Employment Outcomes of Individuals With ID/DD
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Virginia Commonwealth University (Other)
Collaborators: National Institute on Disability, Independent Living, and Rehabilitation Research (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: HM20029287
Record Dates: First submitted 2024-08-26; First posted 2024-09-19 (Actual); Last update posted 2025-07-31 (Actual); Status verified 2025-07

CONDITIONS: Intellectual Disability; Developmental Disability
Keywords: Employment Specialist; Job Coaches
MeSH Terms: conditions — Intellectual Disability; Developmental Disabilities

STUDY DESIGN:
Intervention Model Description: The proposed study will be a randomized control trial, participants will be recruited for the study and once consented they will be randomly assigned to the Control group which entails accessing the current VCU-RRTC online course or the intervention group which will receive the VCU-RRTC course plus TA. TA activities and outlines are attached. Participants who are assigned to the control group will have the opportunity to opt in to the TA sessions after the completion of the third data collection time period. The decision to use an RCT is a natural evolution of the initial two phases of the study and will help provide a comparison of the impact and benefit of additional TA. The addition of the additional two measures that will ask participants to self-report on their employment skills and employment outcomes will also provide important information for future studies.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control Group (Placebo Comparator): The current VCU-RRTC online course. Association of Community Rehabilitation Educators, accrediting body that has developed competencies for job coaches and that approved the online curriculum that has been provided through the VCU-RRTC for over a decade.
  Interventions: Other: VCU-RRTC Online Course
- Experimental (Experimental): The VCU-RRTC course plus TA (Technical Assistance). Association of Community Rehabilitation Educators, accrediting body that has developed competencies for job coaches and that approved the online curriculum that has been provided through the VCU-RRTC for over a decade.
  Interventions: Other: VCU-RRTC Online Course; Other: Zoom Technical Assistance Sessions (6 total)

INTERVENTIONS:
Other: VCU-RRTC Online Course — Approved by ACRE as its accrediting body and has been offered virtually through the VCU RRTC for over 15 years. The course currently entails:
  i. Six modules ii. Six online discussion boards iii. Assignments in each module iv. One quiz per module v. Final assignment
Other: Zoom Technical Assistance Sessions (6 total) — Technical Assistance sessions will be provided to small groups of participants of 5-7 via Zoom technology. There will be one virtual TA session for each of the six modules that will last for 1 hour. The TA sessions will be provided by a trained SE expert/ mentor. The TA sessions will have instructional plans so that they are delivered consistently and will align with the associated module's content and will entail application and discussion that facilitates implementation and reflection of the material.
  Arms: Experimental

SUMMARY:
Currently, there are no national pre-requisites for training to become or to be hired as an ES (Employment Specialist). Staff providing employment services have a broad range of educational and training backgrounds. Some individuals have a masters and have completed an ACRE approved course to earn a ACRE (Association of Community Rehabilitation Educators) Basic Employment Certificate in Employment Services while others may have a high school diploma and have not received any additional training. The first phases of the study were important in identifying if the currently identified ACRE competencies are relevant and if the ACRE approved online training course does impact knowledge.

DETAILED DESCRIPTION:
The final phase of the study aims to identify if the addition of technical assistance to the current course not only impacts knowledge of participants but also their self-reported engagement in skills that are outputs of their knowledge acquisition. Additionally, the third phase will link participation in the course and TA (technical assistance) to employment outcomes of individuals with ID/DD (individuals with intellectual and/or developmental disability). These additions address large gaps in the extant literature and research on employment specialists, training, and its impact on employment outcomes.

While, evidence-based practices in SE (Supported Employment) exist, research indicates that these practices are not often put into practice. Furthermore, of the few studies that have explored ES(Employment Specialist) training and its effectiveness, very few have identified if training impacts the employment outcomes of individuals with disabilities. Employment specialists and their skill directly impact the successful employment of individuals with ID/DD. Despite the introduction of SE into the field over four decades ago as well as legislative support, employment outcomes of individuals with remain dismally low. It is necessary to begin to gather evidence of the impact of training as well as feasibility and dosage in order to identify how to prepare employment service providers to better support individuals with disabilities to access employment.

ELIGIBILITY:
Inclusion Criteria:

* Use the VCU RRTC listserv
* Residing or working in the United States
* 18 and older
* have not participated in ACRe training
* Currently providing or will be providing employment services to individuals with ID/DD

Exclusion Criteria:

* Unable to consent
* Under 18
* Pregnant women
* Prisoners

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2024-06-03 (Actual); Primary Completion 2025-04-07 (Actual); Study Completion 2025-04-07 (Actual)

PRIMARY OUTCOMES:
Impact of VCU ACRE on skills and knowledge | after study completed-9 months
  Identify if VCU ACRE Online Course impact skills and knowledge of employment profession The VCU Supported Employment Online Course is designed to provide knowledge and skill development in competitive integrated employment to include supported and customized employment.
  The 40-hour training is presented in six modules. Each module is posted for two weeks for a total of twelve weeks. Course content is delivered through an online course format with recorded audio and video presentations, required reading, practical activities, and online discussions covering the following topics:
  Module 1: Overview and Introduction to Employment First Module 2: Customer Profile and Discovery Module 3: Marketing and Job Development Module 4: Customized Employment Module 5: Job Site Supports Module 6: Social Security and Other Special Topics

SECONDARY OUTCOMES:
Impact of VCU ACRE course plus technical assistance | after study completed-9 months
  The VCU Supported Employment Online Course is designed to provide knowledge and skill development in competitive integrated employment to include supported and customized employment.
  Identify if VCU ACRE Online Course plus technical assistance impact skills and knowledge of employment profession. The 40-hour training is presented in six modules. Each module is posted for two weeks for a total of twelve weeks. Course content is delivered through an online course format with recorded audio and video presentations, required reading, practical activities, and online discussions covering the following topics:
  Module 1: Overview and Introduction to Employment First Module 2: Customer Profile and Discovery Module 3: Marketing and Job Development Module 4: Customized Employment Module 5: Job Site Supports Module 6: Social Security and Other Special Topics

CONTACTS AND LOCATIONS:
Overall Officials: Whitney Ham, Principal Investigator — Virginia Commonwealth University
Locations (1):
- Virginia Commonwealth University, Richmond, Virginia, United States